CLINICAL TRIAL: NCT05438550
Title: 14-day High-dose Tegoprazan Double Therapy Versus Bismuth Quadruple Therapy in First-line Treatment of Helicobacter Pylori Infection: a Prospective, Randomized, Controlled Study
Brief Title: 14-day Double Therapy Versus Bismuth Quadruple Therapy in First-line Treatment of Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, doctoral supervisor of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022SDU-QILU-G003
Record Dates: First submitted 2022-06-20; First posted 2022-06-30 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori Infection; High dose dual therapy; Bismuth-containing quadruple therapy
MeSH Terms: interventions — tegoprazan; BID protein, human; Amoxicillin

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14-day bismuth-containing quadruple therapy (BQT) (Active Comparator): 14-day bismuth-containing quadruple therapy (BQT) Nexium (Esomeprazole, Astrazeneca Pharmaceutical Co., LTD.) 20mg bid Amoxicillin (Amoxicillin, United Laboratories Co., LTD) 1000mg bid Tetracycline (Huanan Brand, Guangdong Huanan Pharmaceutical Co. LTD.) 500mg qid Bismuth potassium Citrate (Lizhu Delle, Lizhu Group Pharmaceutical Factory) 2g bid
  Interventions: Drug: 14-day high-dose Tegoprazan Dual Therapy (HDDT)
- 14-day Tegoprazan high-dose dual therapy (HDDT) (Experimental): 14-day Tegoprazan high-dose dual therapy (HDDT) Tegoprazan（Luo Xin Pharmaceutical Group Co. LTD）50mg bid Amoxicillin (Amoxicillin, United Laboratories Co. LTD) 750mg qid
  Interventions: Drug: 14-day high-dose Tegoprazan Dual Therapy (HDDT)

INTERVENTIONS:
Drug: 14-day high-dose Tegoprazan Dual Therapy (HDDT) — 14-day Tegoprazan high-dose dual therapy (HDDT) Tegoprazan（Luo Xin Pharmaceutical Group Co. LTD）50mg bid Amoxicillin (Amoxicillin, United Laboratories Co. LTD) 750mg qid To investigate the efficacy of high-dose dual therapy of Tegoprazan, a novel p-CAB acid suppressant, combined with amoxicillin for the eradication of Helicobacter pylori
  Other Names: Tegoprazan (Rosin Pharmaceutical Group Co. LTD.) 50mg bid; Amoxicillin (Amoxicillin, United Laboratories Co. LTD) 750mg qid

SUMMARY:
The researchers collected untreated H. pylori positive patients from outpatient clinics. Subjects were randomized to 14 days of dual therapy with Tegoprazan or 14 days of quadruple therapy with bismuth for eradication. At 6 weeks after treatment, subjects underwent another 13C-urea breath test. The eradication rate, adverse reaction rate and patient compliance were calculated.

DETAILED DESCRIPTION:
1. Informed consent: Patients with positive Helicobacter pylori were collected in the outpatient department, and the subjects receiving initial treatment signed informed consent.
2. Safety evaluation: C13 urea breath test, blood routine test, urine routine test, electrolyte test and liver and kidney function test were performed to confirm helicobacter pylori infection.
3. Confirm the inclusion of patients: fill in the case report form and enter group A or group B according to the randomization results.

   Group A: 14-day Tegoprazan high-dose dual therapy (HDDT) Tegoprazan 50mg bid Amoxicillin 750mg qid Group B: 14-day bismuth-containing quadruple therapy (BQT) Esomeprazole 20mg bid Amoxicillin 1000mg bid Tetracycline 500mg qid Potassium bismuth citrate 2g bid
4. Supervised medication: follow up the medication situation and adverse reactions by telephone 14 days after taking medication, and remind the reexamination 6 weeks after stopping medication.
5. Results: C13 urea breath test was repeated 6 weeks after drug withdrawal. Blood routine, urine routine, electrolytes and liver and kidney function tests were performed.
6. Complete the Case Report Form: Fill in the case report form accurately.
7. Data analysis: SPSS software was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infection (either positive for Helicobacter pylori culture, histopathological test, rapid urease test, C13/C14 urea breath test, or helicobacter pylori antigen test in feces).
* Patients who have not previously received helicobacter pylori eradication therapy.

Exclusion Criteria:

* Serious underlying diseases, such as liver insufficiency, renal insufficiency, immunosuppression, malignant tumor, coronary heart disease (angina pectoris or coronary artery stenosis ≥ 75%).
* Those who are not willing to take contraceptive measures during pregnancy, lactation or the trial.
* Active gastrointestinal bleeding.
* History of drug allergy.
* Medication history of bismuth, antibiotics and PPI within 4 weeks.
* Other behaviors that may increase the risk, such as alcohol and drug abuse.
* Unable or unwilling to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-02-14 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | immediately after the procedure
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | Immediately after the procedure
  Rate of adverse reactions
Patient compliance | Immediately after the procedure
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China